CLINICAL TRIAL: NCT00126204
Title: Adjunctive Treatment With Doxycycline in Endovascular Aneurysm Repair
Brief Title: Adjunctive Treatment With Doxycycline to Enhance the Durability of Endovascular Aortic Aneurysm Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Foundation for Barnes-Jewish Hospital (Other)
Organization: Barnes-Jewish Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00012-0904-02
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2006-09

CONDITIONS: Aortic Aneurysm
Keywords: endoleak; doxycycline; matrix metalloproteinase; inflammation; endograft; circulating markers
MeSH Terms: conditions — Aortic Aneurysm; Endoleak; Inflammation | interventions — Doxycycline

INTERVENTIONS:
Drug: Doxycycline

SUMMARY:
The durability of endovascular aneurysm repair (EVAR) has been limited by development of endoleaks which may be secondary to progressive aortic degeneration by matrix metalloproteases (MMP). Doxycycline is a known inhibitor of the MMP family of enzymes in aneurysms. The investigators propose a randomized, controlled trial of adjuvant doxycycline therapy with EVAR to determine its effects on re-intervention, aneurysm shrinkage and serum markers of aneurysmal degeneration.

DETAILED DESCRIPTION:
Patients will be consented and enrolled at the time of their clinic visit or admission to the hospital for a planned EVAR, in accordance with institutional review board guidelines. Demographic, risk factor and medication regimen data will be obtained from the patient's clinical chart. Patients will be randomized to doxycycline therapy (100 mg taken twice daily) or a placebo. The patients will receive their first dose of study medication on the day following surgery, and continue the study therapy for 6 months.

Plasma and serum will be obtained at the time of enrollment (baseline), and at each post-operative follow-up visit during the study as outlined above. Aliquots will be stored at -80ºC until assayed. Measurements of the circulating markers will be performed by commercially available assays for plasma MMP-9 (R&D Systems, Minneapolis, MN), serum IL-6 (R&D Systems) , IL-8 (R&D Systems), IFN-gamma (R&D Systems), and CRP (Bio-Check, Burlingame, CA) Data will be collected from the pre-operative and all post-operative CT scans regarding maximal aneurysm diameter and transverse neck diameter at 5 mm, 10 mm and 15 mm below the takeoff of the lowest renal artery. All documented endoleaks and their clinical type will be recorded, as will any re-intervention related to the graft or aneurysm.

The primary end-points of the study related to aneurysm measurements will be an increase or decrease in any of the diameter measurements of the aorta by 2 mm or more on 2 consecutive CT scans or a change of 5 mm or more on any single scan. Of the circulating markers, an additional primary endpoint will be a 50% reduction in baseline MMP-9 after endografting. Secondary endpoints will be significant reductions over baseline in circulating IL-6, IL-8, IFN-γ, and CRP. An a priori power analysis indicates that at 6 months, reductions in circulating levels of these markers by 50% can be detected with a β-error of less than 0.1 and α-error of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an abdominal aortic aneurysm (AAA) with a maximum diameter of > or = 4.5 cm
* Planned aneurysm exclusion with endoluminal stent graft (any brand)

Exclusion Criteria:

* Known malignancy not to include prostate cancer or any history of cancer that has not had a recurrence in the last 5 years.
* Hypersensitivity to doxycycline or any of its components
* Pregnancy
* Ruptured AAA
* Extension of covered portion of the graft above the renal arteries
* Previous endoluminal aneurysm repair

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2004-03; Study Completion 2006-07

PRIMARY OUTCOMES:
Change in aortic measurements by > 2 mm on 2 consecutive scans
Change in aortic measurement by > 5 mm on a single scan
50% reduction in baseline plasma MMP-9 at 6 months

SECONDARY OUTCOMES:
Significant reductions at 6 months in serum interleukin-6 (IL-6)
Significant reductions at 6 months in serum IL-8
Significant reductions at 6 months in serum interferon-gamma
Significant reductions at 6 months in serum C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: John A Curci, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine / Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Result] Hackmann AE, Rubin BG, Sanchez LA, Geraghty PA, Thompson RW, Curci JA. A randomized, placebo-controlled trial of doxycycline after endoluminal aneurysm repair. J Vasc Surg. 2008 Sep;48(3):519-26; discussion 526. doi: 10.1016/j.jvs.2008.03.064. Epub 2008 Jul 15. PMID 18632241